CLINICAL TRIAL: NCT05909566
Title: Respiratory Support and Treatment for Efficient and Cost-Effective Care
Acronym: REST EEC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christopher Horvat (Other)
Collaborators: Beckwith Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Christopher Horvat, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY23010030
Record Dates: First submitted 2023-05-24; First posted 2023-06-18 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Bronchiolitis
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Intervention Model Description: We will be providing clinical decision support tools for children receiving HHFNC for bronchiolitis, testing the impact of decision support compared to usual care in a pragmatic randomized trial. All subjects will receive standard of care.
  Decisions regarding management will be at the discretion of the treating provider and will not be restricted or altered in any way.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- HHFNC + Clinical decision Support (Experimental): Standardized HHFNC weaning coupled with clinical decision support consisting of electronic record embedded reminders to the clinical team to wean HHFNC
  Interventions: Other: Clinical Decision Support (CDS); Device: HHFNC Weaning
- HHFNC Weaning (Active Comparator): Team does not receive clinical decision support reminders to wean the HHFNC
  Interventions: Other: Clinical Decision Support (CDS); Device: HHFNC Weaning

INTERVENTIONS:
Other: Clinical Decision Support (CDS) — Education to front line clinicians and staff on standardized implementation and weaning of HHFNC and standardized assessments of patient work of breathing. HHFNC implementation and weaning strategies will be based on age-specific practices recommended by the American Academy of Pediatrics. Education will be undertaken by dedicated clinical educators.
Device: HHFNC Weaning — Wean patient off oxygen and flow as oxygenation and work of breathing improves.

SUMMARY:
This project aims to answer the essential questions about the management of acute, pediatric respiratory illness, accelerate recovery from these all-too-common diseases, curb unnecessary costs of care, and demonstrate UPMC Children's Hospital of Pittsburgh's capabilities as the premier, world-class leader in the arena of pediatric learning healthcare systems. REST EEC will focus on the question of whether clinical decision support (CDS) facilitates the standardization of the initiation and weaning of heated high flow nasal cannula (HHFNC) for bronchiolitis.REST EEC will focus on whether the application of CDS improves adherence to a standardized guideline and leads to improved patient-centered outcomes.

ELIGIBILITY:
Inclusion Criteria:

* <2 years of age Bronchiolitis WOB Score >2

Exclusion Criteria:

* Immunocompromised
* Immunosuppressed
* Chronic lung disease
* Congenital heart disease with baseline cardiorespiratory manifestations

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 198 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
HFNC duration | Timeframe consists of a start time of either randomization or the last documentation of positive pressure ventilation (whichever is later) and the last documentation of HFNC in the electronic flowsheet, up to 30 days
  Amount of time patient is on HFNC

SECONDARY OUTCOMES:
Respiratory support free days | From date the start of respiratory support until the first documented respiratory support free day, up to 30 days
  Days alive and free of intensive care unit-based respiratory
Hospital length of stay | From date of admission until discharge or date of death from any cause, whichever came first, assessed up to 90 days.
  Days admitted in hospital
Organ support free days | From date of admission until the first day of ICU-based respiratory or cardiovascular organ support or discharge or date of death from any case, whichever came first, assessed up to 30 days
  Days alive and free of ICU-based respiratory or cardiovascular organ support
Time to oral intake | From date of ending HHFNC until first documented oral intake, assessed up to 30 days
  Time from HHFNC and oral intake
Ostensible respiratory distress measured by a respiratory severity score | Through study completion, an average of 1 week
  The product of mean airway pressure and the fraction of inspired oxygen
Cost of hospitalization | Days from admission to discharge from hospital or date of death, up to 90 days. Of note, an earlier outcome was listed for 90-day cost of care and the redundancy with this outcome was recognized, so the 90-day cost of care outcome was removed.
  Totality of expenses incurred by a hospital in providing its services and care
Mortality | From date of admission until death from any cause, assessed up to 90 days
  Patient Death
PICU length of stay | From data of admission to PICU to discharge from the PICU or death from any cause, whichever came first, assessed up to 90 days.
  Days admitted in the PICU. This is added to reconcile the plan to evaluate this outcome and its noted absence from this website, as pointed out by a reviewer while working to publish the trial design.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Horvat, MD, Principal Investigator — UPMC Children's Hospital of Pittsburgh
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Horvat CM, Suresh S, James N, Aneja RK, Au AK, Berry S, Blumer A, Bricker K, Clark RSB, Dolinich H, Hahner S, Jockel C, Kalivoda J, Loar I, Marasco D, Marcinick A, Marroquin O, O'brien J, Pelletier J, Ramgopal S, Venkataraman S, Angus DC, Butler G. A randomized, embedded, pragmatic, Bayesian clinical trial examining clinical decision support for high flow nasal cannula management in children with bronchiolitis: design and statistical analysis plan. Trials. 2024 Jul 16;25(1):484. doi: 10.1186/s13063-024-08327-y. PMID 39014495